CLINICAL TRIAL: NCT06341595
Title: Concurrent Chemoradiotherapy Combined With Sintilimab as Neoadjuvant Therapy for Advanced Gastric Cancer Patients With Para-aortic Lymph Node Metastasis: a Single-arm, Phase II, Exploratory Study.
Brief Title: Concurrent Chemoradiotherapy Combined With Sintilimab as Neoadjuvant Therapy for GC Patients With PALM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123322
Record Dates: First submitted 2023-11-14; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer; Gastric Cancer Metastatic to Regional Lymph Nodes
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy (Experimental): sintilimab combined with chemotherapy and radiotherapy
  Interventions: Drug: Sintilimab; Radiation: Extraperitoneal radiation therapy; Drug: Oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: Sintilimab — Sintilimab: 200mg iv q3w d1, 4-6 cycles
Radiation: Extraperitoneal radiation therapy — Radiotherapy using extraperitoneal radiation therapy, once a day, 5 times a week, 1.8-2 Gy/f, a total of 45-50.4 Gy (lymph node lesion radiation dose of 60-66 Gy)
Drug: Oxaliplatin — oxaliplatin: 130mg/m^2, D1, Q3W, 4-6 cycles
Drug: S-1 — S-1: 40mg/m^2, bid, d1-14, 4-6 cycles

SUMMARY:
This trial is a prospective, single arm, single center, phase II clinical study aimed at subjects with advanced gastric cancer and para aortic lymph node metastasis, exploring the feasibility and safety of Sintilimab Injection combined with synchronous chemo-radiotherapy as neoadjuvant therapy.

Patients will receive sintilimab Injection (200mg iv q3w d1) combined with concurrent radiotherapy and chemotherapy. The chemotherapy regimen will use oxaliplatin 130mg/m2+S-1 40mg/m2 bid d1-14. Radiotherapy is performed using intraperitoneal radiation therapy, once a day, five times a week, at a dose of 1.8-2 Gy/f, for a total of 45-50.4 Gy (60-66 Gy for lymph node lesions). Radiation therapy starts from the second cycle of Sintilimab Injection combined with chemotherapy. The subjects underwent imaging evaluation after completing 4 cycles of combination chemotherapy and radiation therapy with Sintilimab Injection. Evaluated as a surgical subject (surgical conditions: imaging evaluation of enlarged lymph nodes adjacent to the abdominal aorta with PR or no significant activity), radical surgery will be performed within 4 weeks after the last study drug treatment. After surgery, the researcher will determine the necessity of adjuvant treatment and develop an adjuvant treatment plan based on the subject's condition. Subjects evaluated as inoperable will have their best follow-up treatment plan determined by the researcher.

ELIGIBILITY:
Inclusion criteria:

* Able to provide informed consent and willing to sign an approved consent form;
* age ≥ 18 years old and ≤ 75 years old, male and female;
* Has histologically confirmed diagnosis of gastric or GEJ adenocarcinoma;
* patients with advanced gastric cancer who have para aortic lymph node metastasis at the initial treatment and whose primary tumor site can be treated with D2 radical operation;
* peritoneal exploration to exclude peritoneal metastasis, liver metastasis and other metastasis;
* CT or MRI, PET-CT and other examinations suggest that there is only one unresectable factor, namely, para aortic lymph node metastasis;
* has not receive previous anti-tumor treatment (radiotherapy, chemotherapy, targeted or immunotherapy, etc.);
* Has at least one measurable lesion as defined by RECIST 1.1 as determined by investigator assessment.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* expected survival time >3 months;
* sufficient organ function, the subject needs to meet the following laboratory indicators:

  1. The absolute neutrophil count (ANC) ≥ 1.5x109/l without granulocyte colony stimulating factor in the past 14 days.
  2. Platelets ≥ 100 without blood transfusion in recent 14 days × 109/l.
  3. Hemoglobin >9g/dl without blood transfusion or use of erythropoietin in recent 14 days;
  4. Total bilirubin ≤ 1.5 × Upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) were ≤ 2.5 × ULN (ALT or AST ≤ 5 allowed for subjects with liver metastasis × ULN);
  6. Blood creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by Cockcroft Gault formula) ≥ 60 ml/min;
  7. Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
  8. Thyroid function was normal, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at the timing of enrollment. Women of non-childbearing potential was defined as having a cessation of menses for one or more year or having surgical sterilization/Hysterectomy
* Participants of childbearing potential must be willing to use an adequate method of contraception （method with failure rate less than 1% in a year）for the course of the study through 120 days after the last dose of study medication or through 180 days of last dose of chemotherapy.

Exclusion criteria:

* HER-2 positive status
* peritoneal or other organ metastasis;
* endoscopy shows signs of active bleeding, and history of gastrointestinal perforation and /or fistula within 6 months before enrollment.;
* other malignant diseases other than gastric cancer diagnosed within 5 years before the first administration (excluding skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or carcinoma in situ after radical resection);
* Is currently participating in and receiving study therapy , or having been treated with another research drug or with an investigational medical devices within 4 weeks before the first administration;
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, anti-PD L2 , anti-CD137,anti-CTLA-4 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137);
* have received systemic treatment with Chinese patent drugs with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control ascites) within 2 weeks before the first administration;
* active autoimmune disease requiring systemic treatment (such as the use of disease modifying drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments;
* being treated with systemic glucocorticoids (excluding nasal spray, inhalation or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose of the study;

Note: physiological doses of glucocorticoids (≤ 10 mg/ day of prednisone or equivalent) are allowed;

* Known history of allogeneic organ (except corneal transplantation) or allogeneic hemopoietic stem cell transplantation;
* Known allergy or hypersensitivity to the investigational drugs Sintilimab, Oxaliplatin, S-1 or excipients;
* there are many factors that affect oral drugs (such as inability to swallow, after gastrointestinal resection, chronic diarrhea and intestinal obstruction, cardiac and pyloric obstruction affecting eating and gastric emptying);
* have not fully recovered from the toxicity and / or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or reaching baseline, excluding fatigue or hair loss);
* Human Immunodeficiency Virus (HIV) infection (HIV antibody positive) (i.e. HIV 1/2 antibody positive);
* uncontrolled active hepatitis B (defined as HBsAg positive with HBV-DNA copy number greater than the upper limit of normal value in the laboratory of the research center);

Note: hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load was <1000 copies /ml (200 iu/ml) before the first dose, and subjects should receive anti HBV treatment throughout the study drug treatment period to avoid virus reactivation
2. For subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), prophylactic anti HBV treatment is not required, but viral reactivation needs to be closely monitored

   * active HCV infected subjects (HCV antibody positive and HCV-RNA level higher than the lower limit of detection);
   * vaccinated with live vaccine within 30 days before the first administration (cycle 1, day 1);

Note: it is allowed to receive inactivated virus vaccine for injection against seasonal influenza within 30 days before the first administration; However, live attenuated influenza vaccines administered intranasally are not allowed.

* Women who are pregnant or nursing.
* there are any serious or uncontrollable systemic diseases, such as:

  1. The resting ECG has major abnormalities in rhythm, conduction or morphology, and the symptoms are serious and difficult to control, such as complete left bundle branch block, heart block above grade II, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) classification ≥ 2;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before enrollment;
  4. Blood pressure control was not ideal (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
  5. There was a history of non infectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or there was currently clinically active interstitial lung disease;
  6. Active pulmonary tuberculosis;
  7. The presence of active or uncontrolled infections requiring systemic treatment;
  8. There were clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor control of diabetes (fasting blood glucose (FBG) > 10mmol/l);
  11. The urine routine showed that the urine protein was ≥ + +, and the 24-hour urine protein quantitation was confirmed to be > 1.0 G;
  12. Those who have mental disorders and cannot cooperate with treatment;
* Other acute or chronic diseases, mental illness, or abnormal laboratory test results that may lead to the following outcomes: increase the risk of participating in study or study drug administration, or interfere with the interpretation of the study results and considered by investigator as "NOT" eligible to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | 24 months
  Recurrence free survival of patients undergoing surgery after Sintilimab Injection combined with concurrent chemoradiotherapy

SECONDARY OUTCOMES:
R0 resection rate | 12 months
  Proportion of patients with R0 resection who underwent surgery in all enrolled patients.
Objective response rate (ORR) | 24 months
  Proportion of participants in complete and partial remission
Major pathological response rate (MPR) | 12 months
  Proportion of patients with residual survival tumor ≤ 10% in all enrolled patients during surgery
Overall survival (OS) | 24 months
  Median survival time of all subjects from enrollment to death from any cause
Adverse reactions | 24 months
  According to the adverse event data of CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China